CLINICAL TRIAL: NCT01096979
Title: A Double-Masked, Evaluation of the Safety and Efficacy of LIPO-102 for the Reduction of Subcutaneous Abdominal Adiposity
Brief Title: An Evaluation of the Safety and Efficacy of LIPO-102 for the Reduction of Subcutaneous Abdominal Adiposity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-102-CL-04
Record Dates: First submitted 2009-10-16; First posted 2010-03-31 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Subcutaneous Abdominal Adiposity
Keywords: Subcutaneous Adipose Tissue Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LIPO-102, High (Experimental): LIPO-102, High
  Interventions: Drug: LIPO-102
- LIPO-102, Low (Experimental): LIPO-102, Low
  Interventions: Drug: LIPO-102
- Placebo (Experimental): Pbo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-102 — subcutaneous injection
  Arms: LIPO-102, High; LIPO-102, Low
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-masked evaluation of the safety and efficacy of LIPO-102 for the reduction of subcutaneous abdominal adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant female
* Good general health
* Sufficient abdominal fat for injections
* Signed informed consent
* BMI greater than or equal to 18 and less than 28 kg/m2
* History of stable weight in past 3 months

Exclusion Criteria:

* Known hypersensitivity to study drugs
* Treatment with an investigational agent within 30 days of first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks
  Vital signs, injection site assessment, clinical laboratory tests (hematology, serum chemistry, lipid panel including FFA, and urine dipstick analysis) and adverse events.
Reduction in abdominal adiposity | 8 weeks
Waist circumference | 8 weeks

SECONDARY OUTCOMES:
Photographic assessments | 8 weeks
  Abdominal volume reductions
Skin-fold caliper measurements | 8 weeks
Patient and clinician Global Impression of severity survey | 8 weeks
Patient and clinician global impression of change questions | 8 weeks
Abdominal appearance questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anaheim, California
  - San Diego, California